CLINICAL TRIAL: NCT05529810
Title: Characteristics and Consequences of Coronary Angiograms Performed in Intensive Care Patients
Acronym: Coro-ICU
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8639
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Coronary angiography; Cardiogenic shock; Cardio-respiratory arrest
MeSH Terms: conditions — Acute Coronary Syndrome; Shock, Cardiogenic; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary angiography is a key examination in the management of many patients hospitalized in intensive care units. The most frequent indication remains the performance of a gesture of unblocking of part of the coronary network in the context of an acute coronary syndrome (ACS) complicated by cardiogenic shock (CS) and/or cardiac arrest. cardio-respiratory (ACR). However, there are other indications in intensive care, in particular for diagnostic purposes. Given the lack of harmlessness of this procedure in itself and the consequences of intra-hospital transport outside intensive care units for patients who are sometimes very unstable, the risk-benefit balance before performing a coronary angiography requires always be properly assessed by the resuscitating physician.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Patients hospitalized in Intensive Medicine - Resuscitation between January 1, 2015 and January 1, 2020 in whom a coronary angiography was performed.
* Patient not objecting to the reuse of their data for scientific research purposes.

Exclusion criteria:

• Patient who has expressed his opposition to the reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) hospitalized in Intensive Medicine - Resuscitation between January 1, 2015 and January 1, 2020 in whom a coronary angiography was performed.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Number of complications occurring in the 3 days following the performance of a coronary angiography during their stay in the intensive care unit | 3 days following the performance of a coronary angiography during their stay in the intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive - Réanimation - CHU de Strasbourg - France, Strasbourg, France